CLINICAL TRIAL: NCT00621699
Title: Pharmacokinetic Drug Interaction Between Ezetimibe and Tacrolimus After Single Dose Administration in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Responsible Party: Prof. Dr. W. Siegmund, MD, Department of Clinical Pharmacology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Eze-Tacro; 2006-006549-14
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Last update posted 2008-02-22 (Estimated); Status verified 2008-02

CONDITIONS: Pharmacokinetics; Drug Interactions; Hypercholesterolemia; Immunosuppression
Keywords: pharmacokinetics; drug interactions; ezetimibe; tacrolimus; human experimentation
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- C (Experimental): administration of 1 tablet Ezetrol(R) (10 mg ezetimibe) and 1 capsule Prograf(R) (5 mg tacrolimus)
  Interventions: Drug: 1 tablet Ezetrol(R) + 1 capsules Prograf(R)
- A (Active Comparator): administration of 1 tablet Ezetrol(R) (10 mg ezetimibe)
  Interventions: Drug: 1 tablet Ezetrol(R) (ezetimibe), MSD Sharp & Dohme GmbH, Germany
- B (Active Comparator): administration of 1 capsule Prograf(R) (5 mg tacrolimus)
  Interventions: Drug: 1 capsule Prograf(R) (tacrolimus), Astellas Pharma GmbH, Germany

INTERVENTIONS:
Drug: 1 tablet Ezetrol(R) (ezetimibe), MSD Sharp & Dohme GmbH, Germany — administration of 1 tablet Ezetrol(R) (10 mg ezetimibe), 0-144 h blood sampling, 0-5 d urine sampling (24 h intervals) and 0-10 d feces sampling
  Other Names: Ezetrol
  Arms: A
Drug: 1 capsule Prograf(R) (tacrolimus), Astellas Pharma GmbH, Germany — administration of 1 capsule Prograf(R) (5 mg tacrolimus), 0-144 h blood sampling
  Other Names: Prograf
  Arms: B
Drug: 1 tablet Ezetrol(R) + 1 capsules Prograf(R) — administration of 1 tablet Ezetrol(R) (10 mg ezetimibe) and 1 capsule Prograf(R) (5 mg Tacrolimus), 0-144 h blood sampling, 0-5 d urine sampling (24 h intervals) and 0-10 d feces sampling
  Other Names: Ezetrol+Prograf
  Arms: C

SUMMARY:
The purpose of this study is to confirm a significant influence of ezetimibe and tacrolimus on each others pharmacokinetics

DETAILED DESCRIPTION:
Hypercholesterolemia is a frequent finding in organ transplant recipients receiving immunosuppressive drugs such as tacrolimus. To prevent increased cardiovascular morbidity and mortality in these patients, co-medication with lipid-lowering statins is recommended. However, treatment with statins is limited in many patients by insufficient cholesterol-lowering efficacy, drug interactions and serious adverse drug reactions (e.g. rhabdomyolysis). These patients may benefit from comedication with the cholesterol absorption inhibitor ezetimibe. Since tacrolimus and ezetimibe were shown to be substrates of the efflux transporter ABCB1 (P-glycoprotein), drug interactions between both compounds may occur. Therefore, this clinical study in healthy subjects was initiated to evaluate the clinical relevance of drug/drug interactions between tacrolimus and ezetimibe according to the accepted bioequivalence approach.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 - 45 years
* sex: male and female
* ethnic origin: Caucasian
* body weight: 19 kg/m² to 27 kg/m²
* good health as evidenced by the results of the clinical examination, ECG, and the laboratory check-up, which are judged by the clinical investigator not to differ in a clinical relevant way from the normal state
* written informed consent

Exclusion Criteria:

* known allergy to macrolide antibiotics
* existing cardiac or hematological diseases and/or pathological findings which might interfere with safety, pharmacodynamic effect and/or pharmacokinetics of ezetimibe and sirolimus
* existing hepatic and renal diseases and/or pathological findings which might interfere with safety, pharmacodynamic effect and/or pharmacokinetics of ezetimibe and sirolimus
* existing gastrointestinal diseases and/or pathological findings which might interfere with safety, pharmacodynamic effect and/or pharmacokinetics of ezetimibe and sirolimus
* acute or chronic diseases which could affect drug absorption or metabolism
* history of any serious psychological disorder
* drug or alcohol dependence
* positive drug or alcohol screening
* smokers of 10 or more cigarettes per day
* positive screening results for HIV, HBV and HCV
* volunteers who are on a diet which could affect the pharmacokinetics of the drug
* heavy tea or coffee drinkers (more than 1L per day)
* lactation and pregnancy test positive or not performed
* volunteers suspected or known not to follow instructions
* volunteers who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to as a result of their participation in the study
* volunteers liable to orthostatic dysregulation, fainting, or blackouts
* blood donation or other blood loss of more than 400 ml within the last 12 weeks prior to the start of the study
* participation in a clinical trial during the last 3 months prior to the start of the study
* less than 14 days after last acute disease
* any systemically available medication within 4 weeks prior to the intended first administration unless, because of the terminal elimination half-life, complete elimination from the body can be assumed for the drug and/or its primary metabolites (except oral contraceptives)
* repeated use of drugs during the last 4 weeks prior to the intended first administration, which can influence hepatic biotransformation (e.g. barbiturates, cimetidine, phenytoin, rifampicin)
* repeated use of drugs during the last 2 weeks prior to the intended first administration which affect absorption (e.g. laxatives, metoclopramide, loperamide, antacids, H2-receptor antagonists)
* intake of grapefruit containing food or beverages within 7 days prior to administration
* known allergic reactions to the active ingredients used or to constituents of the pharmaceutical preparation
* subjects with severe allergies or multiple drug allergies

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-09; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Primary characteristics: for ezetimibe: AUC0-∞, Cmax; for tacrolimus: AUC0-∞, Cmax | September 2007 to November 2007

SECONDARY OUTCOMES:
Second. characteristics: for ezetimibe: CLR, Ae (urine), Ae (feces); for ezetimibe glucuronide: AUC0-∞, Cmax, Ae (urine), Ae (feces); for ezetimibe, ezetimibe glucuronide and tacrolimus: AUC0-t, t½, tmax | September 2007 to November 2007

CONTACTS AND LOCATIONS:
Overall Officials: Werner Siegmund, Prof, Principal Investigator — Department of Clinical Pharmacology
Locations (1):
- Department of Clinical Pharmacology, Greifswald, Germany